CLINICAL TRIAL: NCT04754191
Title: A Phase 2 Umbrella Protocol of Enfortumab Vedotin as Monotherapy and Combined With Other Agents in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Enfortumab Vedotin as Monotherapy in Patients With Metastatic Castration-Resistant Prostate Cancer
Acronym: ENCORE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI137651
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: all patients (Experimental): Enfortumab will be administered in monotherapy on days 1, 8, and 15 as part of a 28-day cycle at 1.25 mg/kg up to 125 mg.
  Interventions: Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: Enfortumab vedotin — Cohort A will be treated with enfortumab vedotin on a 28 day cycle for up to 12 months.

SUMMARY:
This is an open-label, phase II umbrella trial assessing the anti-tumor activity of enfortumab alone and in combination with other anti-cancer agents in subjects with metastatic castration-resistant prostate cancer. The trial will open to enrollment in Cohort A, enfortumab monotherapy. Additional cohorts may be added as new drug combinations are identified.

ELIGIBILITY:
Inclusion Criteria:

* Male subject aged ≥ 18 years.
* Histologically or cytologically confirmed adenocarcinoma of the prostate without small cell histology.
* Diagnosis of metastatic or locally advanced, inoperable disease that cannot be treated with definitive intent
* Castrate levels of testosterone as defined as < 50 ng/dL (1.73 nmol/L).
* Prior treatment with at least three or more cycles of taxane therapy (docetaxel or cabazitaxel).

Note: Docetaxel in the newly diagnosed metastatic setting and docetaxel rechallenge allowed.

* Prior treatment with at least one prior Novel Hormone Therapy (NHT), defined as second-generation antiandrogen therapies that include but are not limited to abiraterone acetate, enzalutamide, apalutamide, and darolutamide.
* Subject has received or refused therapies which have shown to improve overall survival and are recommended per National Comprehensive Cancer Network (NCCN) guidelines prior to enrollment in trial. Such agents include but are not limited to docetaxel, cabazitaxel, sipuleucel-T, olaparib, rucaparib, radium-223 and lutetium (177Lu) vipivotide tetraxetan depending on patient eligibility.
* Had disease progression on or after NHT prior to enrolling in the study.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Adequate organ function as defined as:

  * Hematologic:

    * White blood cell count (WBC) ≥ 2000/mm3
    * Absolute neutrophil count (ANC) ≥ 1500/mm3
    * Platelet count ≥ 100,000/mm3
    * Hemoglobin ≥ 9g/dL
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN) unless there is a known history of Gilbert's syndrome.
    * Aspartate aminotransferase (AST)(SGOT)/Alanine aminotransferase (ALT)(SGPT) ≤ 5 × institutional ULN
  * Renal:

    * Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula:
* Highly effective contraception throughout the study as described in Section 7.4.
* Discontinued all previous treatments for cancer (except androgen-deprivation therapy and bone loss prevention treatment) 28 days prior to starting study therapy.
* Recovery to baseline or ≤ Grade 1 CTCAE v 5.0 from toxicities related to any prior treatments, unless Adverse Event(s) (AE(s)) are clinically non-significant and/or stable on supportive therapy as determined by the treating physician.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Prior or concurrent malignancy (other than adenocarcinoma of the prostate). Note: Patients with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial as approved by the Principal Investigator.
* The subject has an uncontrolled, significant intercurrent or recent illness that would preclude safe study participation.
* Clinically significant cardiovascular disease: myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (> New York Heart Association Classification Class IIB) or a serious cardiac arrhythmia requiring medication.
* Known HIV infection with a detectable viral load at the time of screening. Note: Patients on effective antiretroviral therapy with an undetectable viral load at the time of screening are eligible for this trial.
* Known chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection with a detectable viral load.

Note: Patients with an undetectable HBV viral load are eligible. Patients with an undetectable HCV viral load are eligible.

* Live attenuated vaccinations within ≤ 4 weeks of the first study therapy and while on trial is prohibited.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.3. A washout period of prohibited medications for a period of at least 5 half-lives or as clinically indicated should occur prior to the start of treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Proportion subjects achieving a protocol-defined response (as defined below): | 12 months
  To assess the anti-tumor action of the study therapy in subjects with metastatic castrate-resistant prostate cancer, as represented by the proportion of subjects achieving one of the following outcomes:
  Objective response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; Confirmed conversion of circulating tumor cell count (CTC) to <5/7.5 mL blood; Prostate Specific Antigen (PSA) decline ≥ 50% from baseline; or Stable disease ≥ 6 months per Prostate Cancer Working Group 3 (PCWG3)-modified RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Umang Swami, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No